CLINICAL TRIAL: NCT03274700
Title: The Use of Tamsulosin in Treatment of (10-15 mm) Lower Ureteric Stones in Adults With Non-emergent Symptoms: A Prospective Randomized Study
Brief Title: The Use of Tamsulosin in Treatment of (10-15 mm) Lower Ureteric Stones in Adults With Non-emergent Symptoms
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mahmoud eldardery, resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: tamsulosin in ureteric stones
Record Dates: First submitted 2017-08-27; First posted 2017-09-07 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-08

CONDITIONS: Ureteric Stone
MeSH Terms: conditions — Ureterolithiasis | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Patients receive tamsulosin (Active Comparator): Patients who will receive tamsulosin as a treatment for lower ureteric stones from (10-15)mm up to 8 weeks duration.e foll The cases will be followed up as thowing:
  In the first month: abdominal ultrasonography every week, KUB abdomen and pelvis for radiopaque stones.
  At the end of the second month: abdominal ultrasonography, KUB abdomen and pelvis for radiopaque stones.
  At the end of the third month: abdominal ultrasonography, KUB abdomen and pelvis for radiopaque stones, MSCT abdomen and pelvis for radiolucent stones.
  Interventions: Drug: Tamsulosin.
- Patients receive placebo. (Placebo Comparator): Patients who will receive placebo up to 8 weeks duration.The cases will be followed up as following:
  In the first month: abdominal ultrasonography every week, KUB abdomen and pelvis for radiopaque stones.
  At the end of the second month: abdominal ultrasonography, KUB abdomen and pelvis for radiopaque stones.
  At the end of the third month: abdominal ultrasonography, KUB abdomen and pelvis for radiopaque stones, MSCT abdomen and pelvis for radiolucent stones.
  Interventions: Drug: Placebo.

INTERVENTIONS:
Drug: Tamsulosin. — Patients who will receive tamsulosin as a treatment for lower ureteric stones from (10-15)mm up to 8 weeks duration.
  Arms: Group 1: Patients receive tamsulosin
Drug: Placebo. — Patients who will receive as placebo a treatment for lower ureteric stones from (10-15)mm up to 8 weeks duration.
  Arms: Patients receive placebo.

SUMMARY:
To estimate the efficacy of tamsulosin in:

A - Expulsion of lower ureteric stones from10-15 mm diameters (primary goal).

B - Pain relief and hyronephrosis improvement (secondary goal).

DETAILED DESCRIPTION:
Urolithiasis affects 4-15% of world population and the incidence of this disease is increasing day by day . Of all the urinary tract stones, 20% are ureteral stones, and 70% of these ureteral stones are found in the distal part of the ureters . The goal of treatment of patients suffering from ureteral calculi is to achieve complete stone clearance with minimal morbidity .

Ureteral calculi of any size may be associated with renal obstruction and care must be taken to prevent irreversible damage to kidney, whether patient selects expectant or active treatment . An expectant treatment or watchful waiting approach may be expected to produce spontaneous stone expulsion up to 50% of cases but some complications such as urinary infection, hydronephrosis, and repetitive colicky pain may occur . Once a conservative approach proves to be unsuccessful, interventional treatment becomes necessary. After a period of conservative treatment, however, intervention is often inefficient or has a higher risk for complications due to stone impaction and the associated inflammatory reaction of the ureter . Non-invasive treatment with extracorporeal shockwave lithotripsy and minimal invasive approach with ureteroscopy allow ureterolithiasis to resolve in almost all cases but these procedures are not risk free and they require some experience and not cost effective .

The therapeutic potential of α-blockers for ureteral stone disease has been investigated, prompted by the detection of α-receptors in ureteral smooth muscle cells . We choose to focus on tamsulosin because it is the most frequently studied α-blocker, recommended in urology treatment guidelines, and, in our experience, the most common medical expulsive therapy used by emergency physicians .

The objective of this trial was to evaluate the efficacy of MET with tamsulosin for ureteral stones from 10-15 mm diameter in a randomised, placebo-controlled setting.

ELIGIBILITY:
Inclusion Criteria:

1. Lower ureteric stones from(10-15) mm diameters.
2. Age group equal or more than 18 years.
3. Normal renal function.

Exclusion Criteria:

1. Lower ureteric stones less than 10mm and more than 15 mm diameters.
2. Age group less than 18 years.
3. Associated ureteric strictures.
4. Febrile urinary tract infections.
5. Severe hydronephrosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Theraputic effect of tamsulosin as assessed by number of cases of expulsed ureteric stones. | 1year
  Patients who will receive tamsulosin as a treatment for lower ureteric stones from (10-15)mm up to 8 weeks duration.e foll The cases will be followed up as thowing:
  In the first month: abdominal ultrasonography every week, KUB abdomen and pelvis for radiopaque stones.
  At the end of the second month: abdominal ultrasonography, KUB abdomen and pelvis for radiopaque stones.
  At the end of the third month: abdominal ultrasonography, KUB abdomen and pelvis for radiopaque stones, MSCT abdomen and pelvis for radiolucent stones.

REFERENCES:
- [Background] Pearle MS. Efficacy of tamsulosin in the medical management of juxtavesical ureteral stones. Int Braz J Urol. 2004 Nov-Dec;30(6):546-547. No abstract available. PMID 15748331
- [Background] Wang RC, Smith-Bindman R, Whitaker E, Neilson J, Allen IE, Stoller ML, Fahimi J. Effect of Tamsulosin on Stone Passage for Ureteral Stones: A Systematic Review and Meta-analysis. Ann Emerg Med. 2017 Mar;69(3):353-361.e3. doi: 10.1016/j.annemergmed.2016.06.044. Epub 2016 Sep 8. PMID 27616037
- [Background] Yilmaz E, Batislam E, Basar MM, Tuglu D, Ferhat M, Basar H. The comparison and efficacy of 3 different alpha1-adrenergic blockers for distal ureteral stones. J Urol. 2005 Jun;173(6):2010-2. doi: 10.1097/01.ju.0000158453.60029.0a. PMID 15879806